CLINICAL TRIAL: NCT01964534
Title: Randomized Phase II Study of Weekly ABI-007 Plus Gemcitabine or Simplified LV5FU2 as First-line Therapy in Patients With Metastatic Pancreatic Cancer
Brief Title: Efficacy of ABI-007 Plus Gemcitabine or sLV5FU2 as First-line Therapy in Patients With Metastatic Pancreatic Cancer
Acronym: AFUGEM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFUGEM D12-2; 2013-001463-23 (EudraCT Number)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic; Pancreatic; Cancer; Pancreas; GERCOR; Gemcitabine; LV5FU2; ABI-007; PACLITAXEL ALBUMIN-BOUND PARTICLES
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM 1 ABI-007 + Gemcitabine (Active Comparator): ABI-007 : 125mg/m² IV / 30min (day 1, day 8, day 15) Gemcitabine : 1000mg/m² IV /30 min (day 1, day 8, day 15) One cycle every four weeks treatment until progression or limiting toxicity
  Interventions: Drug: ABI-007; Drug: Gemcitabine
- Arm 2 ABI-007 + simplified LV5FU2 (Experimental): ABI-007 : 125mg/m² IV /30 min (day 1, day 15) folinic acid : 400mg/m² IV /2h (day 1, day 15) Bolus 5-FU : 400mg/m² IV /15min 5-FU infusion : 2400mg/m² IV / 46h (day 1-2, day 15-16) One cycle every four weeks Treatment until progression or limiting toxicity
  Interventions: Drug: ABI-007; Drug: simplified LV5FU2

INTERVENTIONS:
Drug: ABI-007 — ABI-007 : 125 mg/m² IV /30min (day 1, day 8, day 15)
  Other Names: Abraxane
Drug: Gemcitabine — 1000 mg/m² IV /30min (day 1, day 8, day 15)
  Other Names: Gemzar
  Arms: ARM 1 ABI-007 + Gemcitabine
Drug: simplified LV5FU2 — Folinic acid: 400 mg/m² IV /2h (day 1, day 15) Bolus 5-FU: 400 mg/m² IV /15min (day 1, day 15) 5-FU infusion: 2400 mg/m² IV /46h (day 1-2, day 15-16)
  Arms: Arm 2 ABI-007 + simplified LV5FU2

SUMMARY:
To evaluate the combination of ABI-007 with gemcitabine or with LV5FU2.

DETAILED DESCRIPTION:
Gemcitabine alone or the triplet combination of 5FU, irinotecan and oxaliplatin (FOLFIRINOX)are the reference 1st line treatment for metastatic pancreatic cancer.

The aim of the AFUGEM study is to evaluate the efficacy of weekly ABI-007 in combination with weekly gemcitabine or with fortnightly simplified LV5FU2 regimen in terms of progression-free survival in patients with previously untreated metastatic pancreatic cancer.

ABI-007 has been approved for commercialization in 38 countries, including the US, Canada, the EU, Australia, China, India and Korea for the treatment of women with metastatic breast cancer. ABI-007 alone and in combination is being evaluated in a number of cancers, including metastatic melanoma, non-small cell lung cancer, pancreatic cancer, and other solid tumors. Conditions which are responsive to paclitaxel such as non-hematological solid tumor malignancies are good clinical candidates for treatment with ABI-007.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically or cytologically proven adenocarcinoma of the pancreas,
3. Metastatic disease confirmed (stage IV),
4. No prior therapy for metastatic disease (in case of previous adjuvant therapy, interval from end of chemotherapy and relapse must be >12 months),
5. At least one measurable or evaluable lesion as assessed by CT-scan or MRI (Magnetic Resonance Imaging) according to RECIST v1.1 guidelines,
6. Age ≥18 years,
7. ECOG Performance status (PS) 0-2,
8. Hematological status: neutrophils (ANC) >1.5x109/L; platelets >100x109/L; haemoglobin ≥9g/dL,
9. Adequate renal function: serum creatinine level <150µM,
10. Adequate liver function: AST (SGOT) and ALT (SGPT) ≤2.5xULN (≤5xULN in case of liver metastases)
11. Total bilirubin ≤1.5 x ULN, albumin ≥25g/L
12. Baseline evaluations performed before randomization: clinical and blood evaluations no more than 2 weeks (14 days) prior to randomization, tumor assessment (CT-scan or MRI, evaluation of non-measurable lesions) no more than 3 weeks (21 days) prior to randomization,
13. Female patients must be surgically sterile, or be postmenopausal, or must commit to using reliable and appropriate methods of contraception during the study and during at least six months after the end of study treatment (when applicable). All female patients with reproductive potential must have a negative pregnancy test (β HCG) within 72 hours prior to starting ABI-007 treatment. Breastfeeding is not allowed. Male patients must agree to use effective contraception in addition to having their partner use a contraceptive method as well during the trial and during at least six months after the end of the study treatment,
14. Registration in a national health care system (CMU included for France).

Exclusion Criteria:

1. History or evidence upon physical examination of CNS metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy)
2. Local or locally advanced disease (stage I to III),
3. Patient uses warfarin,
4. Uncontrolled hypercalcemia,
5. Pre-existing permanent neuropathy (NCI grade ≥2),
6. Known dihydropyrimidine dehydrogenase (DPD) deficiency,
7. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
8. Treatment with any other investigational medicinal product within 28 days prior to study entry,
9. Other serious and uncontrolled non-malignant disease (eg. active infection requiring systemic therapy, coronary stenting or myocardial infarction or stroke in the past 6 months),
10. Known or historical active infection with HIV, or known active infection untreated with hepatitis B or hepatitis C.
11. History or active interstitial lung disease (ILD),
12. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
13. Patients with known allergy to any excipient of study drugs,
14. Concomitant administration of live, attenuated virus vaccine such as yellow fever vaccine and concomitant administration of prophylactic phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | time interval from randomization to the date of first documented disease progression or death from any cause, whichever occurs first.Assessed at 4 months.
  To evaluate the efficacy of weekly ABI-007 in combination with weekly gemcitabine or with fortnightly simplified LV5FU2 regimen in terms of progression-free survival in patients with previously untreated metastatic pancreatic cancer

SECONDARY OUTCOMES:
Tumor Response Rate | Assessed every 2 months during treatment period (- Estimated treatment duration per patient : 6 months).
  Assessed using RECIST version 1.1
Duration of disease control (DDC) | Assessed up to 30 months after the beginning of the study
Overall Survival | time interval from inclusion to the date of death from any cause. Assessed up to 30 months after the beginning of the study.
Quality of life | Assessed from study entry to 1 month after last study drug administration and up to 30 months after the beginning of the study.
  EORTC QLQ C-30
Number of Adverse Events | Assessed from study entry to 1 month after last study drug administration, assessed up to 30 months after the beginning of the study
  To evaluate the safety profile of ABI-007 in combination with sLV5FU2 (NCI CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Bachet, MD, Principal Investigator — Hôpital La Pitié-Salpêtrière
Locations (15):
- France (15):
  - Institut de cancérologie de l'Ouest - Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Hôpital Avicenne, Bobigny
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hôpital Privé Jean Mermoz, Lyon
  - CHU la Timone, Marseille
  - Centre Hospitalier Layné, Mont-de-Marsan
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU de Reims Hôpital Robert Debré, Reims
  - Institut de Cancérologie de l'Ouest - Réné Gauducheau, Saint-Herblain
  - Hôpital Trousseau - CHRU Tours, Tours

REFERENCES:
- [Derived] Bachet JB, Hammel P, Desrame J, Meurisse A, Chibaudel B, Andre T, Debourdeau P, Dauba J, Lecomte T, Seitz JF, Tournigand C, Aparicio T, Meyer VG, Taieb J, Volet J, Monier A, Bonnetain F, Louvet C. Nab-paclitaxel plus either gemcitabine or simplified leucovorin and fluorouracil as first-line therapy for metastatic pancreatic adenocarcinoma (AFUGEM GERCOR): a non-comparative, multicentre, open-label, randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2017 May;2(5):337-346. doi: 10.1016/S2468-1253(17)30046-8. Epub 2017 Feb 28. PMID 28397697
- [Derived] Bachet JB, Chibaudel B, Bonnetain F, Validire P, Hammel P, Andre T, Louvet C; GERCOR group. A randomized phase II study of weekly nab-paclitaxel plus gemcitabine or simplified LV5FU2 as first-line therapy in patients with metastatic pancreatic cancer: the AFUGEM GERCOR trial. BMC Cancer. 2015 Oct 6;15:653. doi: 10.1186/s12885-015-1656-4. PMID 26445094